CLINICAL TRIAL: NCT05891834
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy, Safety, and Pharmacokinetics of 3 Doses of INV-202 With an Optional Open-Label Extension in Patients With Obesity and Metabolic Syndrome
Brief Title: Study of INV-202 in Patients With Obesity and Metabolic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inversago Pharma Inc. (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INV-CL-107
Record Dates: First submitted 2023-05-17; First posted 2023-06-07 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Obesity; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Low dose (Experimental): INV-202, 10 mg
  Interventions: Drug: INV-202
- High dose (Experimental): INV-202, 50 mg
  Interventions: Drug: INV-202
- Placebo (Placebo Comparator): Placebo Matching size and number of tablets
  Interventions: Drug: Placebo
- Middle Dose (Experimental): INV-202, 20 mg
  Interventions: Drug: INV-202

INTERVENTIONS:
Drug: INV-202 — tablet, once daily, oral
  Arms: High dose; Low dose; Middle Dose
Drug: Placebo — tablet, once daily, oral
  Arms: Placebo

SUMMARY:
The study is designed to assess the efficacy, safety, tolerability, and transformation within the human body of INV-202 investigational drug in the treatment of adult participants with obesity and metabolic syndrome.

DETAILED DESCRIPTION:
This will be a 2-part study. Part A will be a randomized, double-blind, placebo-controlled, dose ranging, multicenter study assessing the efficacy, safety, tolerability, and PK of INV-202 for the treatment of adult participants with obesity (BMI 30 kg/m2) and metabolic syndrome.

An informed consent form (ICF) must be signed by the participant before any study-related procedures are performed.

Each participant will be allowed 1 retest during the screening period if they have an abnormal test result not meeting eligibility criteria that is deemed transient by the investigator. Participants who did not meet all eligibility criteria may be re-screened once, with approval of the medical monitor.

Participants will return to the study site at Weeks 4, 8, 12 and 16. At these visits, the same assessment as baseline will be completed.

During Part A, a subset of approximately 20 to 30 participants from an estimated 3 to 4 study sites will have DEXA performed at baseline and Week 16 for exploratory assessments of change in total body fat percentage and skeletal muscle mass. Additional exploratory measures will include lung function with oscillometry. Any participant who withdraws from Part A before completing treatment will be requested to return for an early termination visit, at which time the procedures normally scheduled for the Week 16 visit will be conducted.

Participants completing Part A will be eligible to enroll to the open-label extension (OLE), Part B, if they did not have significant noncompliance with study drug, visits, or procedures, and did not meet any withdrawal criteria. During Part B, the efficacy and safety of INV-202 20 mg daily (pending results of chronic toxicology studies and/or findings from this and other ongoing clinical studies, the alternative dose would be 10 mg) will be further evaluated over an additional 36 weeks, through Week 52.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants from 18 to 75 years of age 2. Able and willing to provide informed consent and to comply with scheduled visits and study procedures 3. BMI ≥ 30 kg/m2 4. Presence of at least 3 of the 5 following criteria at screening: i. Increased waist circumference (males, ≥40 inches; females, ≥35 inches) ii. Fasting glucose ≥ 100 mg/dL in the last 3 months or an HgbA1C > 5.7% iii. Triglycerides ≥ 150 mg/dL or 1.69 mmol/L iv. HDL < 40 mg/dL or 1.03 mmol/L for males or < 50 mg/dL or 1.29 mmol/L for females v. Hypertension (systolic >130 mmHg and/or diastolic > 85 mmHg) or treated for hypertension

Exclusion Criteria:

1. Significant medical condition, that in the opinion of the investigator, will place the participant at risk during the study or that will confound the study endpoints
2. Active substance abuse including inhaled, oral, or injection drugs in the past 12 months
3. Use of cannabis or cannabinoid-containing compounds within 90 days prior to screening
4. Pregnancy, planned pregnancy, potential for pregnancy, breast feeding, or unwillingness to use highly effective birth control during the study
5. History of significant liver disease or evidence of moderate to severe hepatic impairment
6. History of epilepsy or intracranial surgery
7. Diabetes requiring medication for management (a diagnosis of diabetes that is well controlled with diet and exercise is not exclusionary)
8. Bariatric surgery, use of a GLP-1 agonists or other weight-loss drug, or significant weight change (> 5 kg or 11 pounds) in the past 3 months
9. Participants taking any drug that may be used for weight loss (eg, liraglutide, semaglutide, tirzepatide, orlistat sibutramine phenylpropanolamine , mazindol , phentermine alone or in combination with topiramate, lorcaserin , naltrexone in combination with bupropion)
10. Use of systemic corticosteroids (topical and inhaled corticosteroids are not excluded)
11. Participants with an active diagnosis or history of a significant psychiatric disorder, including but not limited to the following:

    Major depression within the last 2 years
    * Any history of a suicide attempt or suicidal ideation
    * A history of other severe psychiatric disorder (eg, schizophrenia, bipolar disorder)
    * Taking any of the following medications: antidepressants, atypical antipsychotics and mood stabilizers such as imipramine, amitriptyline, mirtazapine, paroxetine, phenelzine, chlorpromazine, thioridazine, clozapine, olanzapine, valproic acid, lithium
12. Score on the 9-question Patient Health Questionnaire (PHQ-9) of
13. Current or active malignancy within the past 5 years, except for cancer in situ, or nonmelanoma skin cancer, such as basal cell or squamous cell carcinoma that has been completely resected
14. A history thyroid disease; the only exception would be a participant who has undergone a complete thyroid ablation/resection
15. QTc > 500 ms at baseline
16. Any chronic medications with effects on blood pressure, lipids, or blood glucose started or changed within the past 3 months or at risk of requiring a change during the study
17. Participants taking a strong inducer or inhibitor of cytochrome P450 3A4, 2D6, or 2C19 by screening; these medications are prohibited during the entire duration of the study
18. Having taken any investigational compound within 30 days, or 5 half-lives of the drug, whichever is longer, before the screening visit
19. Previous use of INV-202
20. Participants that, in the opinion of the investigator, are unsuitable for the study or unlikely to comply with all study procedures and treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of INV-202 on body weight loss in participants with obesity and metabolic syndrome | Week 16
  Mean change from baseline in body weight at Week 16 for INV-202 versus placebo

SECONDARY OUTCOMES:
To evaluate the effect of INV-202 on weight (marker of metabolic syndrome) | Week 16
  Mean percent change from baseline at each site visit for the following:
  Percent change in weight
To evaluate the effect of INV-202 on waist circumference (marker of metabolic syndrome) | Week 16
  Mean change from baseline at each site visit for the following:
  Change in waist circumference
To evaluate the effect of INV-202 on lipids (marker of metabolic syndrome) | Week 16
  Mean change from baseline at each site visit for the following:
  Change in lipids (LDL, VLDL, HDL, total cholesterol, ApoB) results by central laboratory testing
To evaluate the effect of INV-202 on glucose control (marker of metabolic syndrome) | Week 16
  Mean change from baseline at each site visit for the following:
  Change in markers of glucose control (HgbA1C) results by central laboratory testing
To evaluate the effect of INV-202 on glucose control (marker of metabolic syndrome) | Week 16
  Mean change from baseline at each site visit for the following:
  Change in markers of glucose control (insulin) results by central laboratory testing
To evaluate the effect of INV-202 on glucose control (marker of metabolic syndrome) | Week 16
  Mean change from baseline at each site visit for the following:
  Change in markers of glucose control (C-peptide) results by central laboratory testing

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (24):
- Canada (24):
  - Office of David H. Shu, MD, New Westminster, British Colombia
  - Centricity Research -New Minas, New Minas, Nova Scotia
  - Aggarwal and Associates, Limited, Brampton, Ontario
  - Wharton Medical Clinic (WMC) - Toronto, Hamilton, Ontario
  - Milestone Research Inc, London, Ontario
  - Centricity Research - Oshawa, Oshawa, Ontario
  - Bluewater Clinical Research Group Inc, Sarnia, Ontario
  - Canadian Phase Onward Inc., Toronto, Ontario
  - Dr. Anil K. Gupta Medicine Professional Corporation, Toronto, Ontario
  - Dr. Sameh Fikry Medicine Professional Corporation, Waterloo, Ontario
  - Clinical Research Solutions, Waterloo, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - DIEX Research Joliette, Joliette, Quebec
  - Centricity Research - Levis, Lévis, Quebec
  - Centricity Research - Mirabel, Mirabel, Quebec
  - 9109-0126 Quebec Inc, Montreal, Quebec
  - Centricity Research - Pointe-Claire, Pointe-Claire, Quebec
  - DIEX Research Quebec, Québec, Quebec
  - Centre des maladies lipidique deq Quebec, CMLQ Inc., Québec, Quebec
  - Alpha Recherche Clinique - Lebourgneuf, Québec, Quebec
  - Alpha Recherche Clinique Val-Bélair, Québec, Quebec
  - Diex Recherche Sherbrooke, Sherbrooke, Quebec
  - Diex Recherche Trois-Rivieres, Trois-Rivières, Quebec
  - Diex Recherche Victoriaville, Victoriaville, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Knop FK, Kunos G, Dicker D, Paquette JS, Aronne L, Frenkel O, Holst-Hansen T, Lalonde K, Lee J, Crater G; trial investigators. Efficacy and safety of monlunabant in adults with obesity and metabolic syndrome: a double-blind, randomised, placebo-controlled, phase 2a trial. Lancet Diabetes Endocrinol. 2025 Nov;13(11):911-923. doi: 10.1016/S2213-8587(25)00216-5. Epub 2025 Sep 29. PMID 41038215